CLINICAL TRIAL: NCT06882291
Title: Intermittent Fasting Diet Versus Resistive Exercise Program on Insulin Resistance in Obese Women With P.C.O.S
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Wesam Samy Elsayed Elmokadem, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005568
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intermittent fasting diet + medical treatment (Experimental): This group will consist of 24 obese PCOS women who will receive a program of Intermittent fasting diet for eight weeks and a medical treatment.
  Interventions: Other: Intermittent fasting diet; Drug: Medical treatment
- Resistive exercise program + medical treatment (Experimental): This group will consist of 24 obese PCOS women who will receive a resistive exercise program for 30 minutes 5 times/week for eight weeks and a medical treatment.
  Interventions: Other: Resistive exercise program; Drug: Medical treatment
- Medical treatment (Active Comparator): This group will consist of 24 obese PCOS women who will receive a medical treatment only.
  Interventions: Drug: Medical treatment

INTERVENTIONS:
Other: Intermittent fasting diet — Women in the first experimental group will follow an intermittent fasting diet, where they eat for 8 hours and fast for 16. They can skip breakfast or have an early dinner. Meals will include 500-800 calories of high-fiber and protein-rich foods. Participants can start with 2-3 fasts per week and increase gradually. They must drink 2-3L of water daily and can consume zero-calorie beverages. Weekly assessments will track progress.
  Arms: Intermittent fasting diet + medical treatment
Other: Resistive exercise program — Women in the second experimental group will receive medical treatment and follow an 8-week resistive exercise program (30 min, 5 days/week). Exercises target the upper body, abdomen, and lower limbs, starting with a 10-min warm-up, followed by 30 min of resistance training (biceps curls, triceps exercises, chest press, plank, crunches, squats, lunges, hamstring, and quadriceps curls), and ending with a 10-min cool-down. Repetitions are logged weekly for assessment.
  Arms: Resistive exercise program + medical treatment
Drug: Medical treatment — Each woman in the three groups will receive medical treatment (metformin tablets) for eight weeks and the dose will prescribed by the gynecologist during the first visit. Patients will be asked to attend the clinic each month for routine monitoring.
  Other Names: Metformin tablets

SUMMARY:
This study will be carried out in an attempt to know which is more effective, Intermittent fasting diet or resistive exercise program on insulin resistance in obese woman with polycystic ovarian syndrome.

DETAILED DESCRIPTION:
Polycystic ovarian syndrome (PCOS) significantly impacts women, since the broad spectrum of clinical manifestations associated with it are significant and include reproductive dysfunction, menstrual irregularities, and an increased risk of infertility. However, the consequences of PCOS go beyond the reproductive axis, with psychological and social impairments, including stress, depression, anxiety and sexual dissatisfaction. There is also a high prevalence of dyslipidemia, hyperinsulinemia, obesity, hypertension, and glucose intolerance which are risk factors that predispose women to cardiovascular disease (CVD) and diabetes mellitus type 2 (DM2).

Improving Insulin resistance and excess adiposity are therefore key targets in PCOS management. International Evidence Based Guideline for the Assessment and Management of PCOS , highlights lifestyle intervention as the primary early management strategy. Lifestyle interventions are traditionally defined as those designed to improve dietary intake or physical activity through appropriate behavioural support. Time restricted eating (TRF), where patients are asked to consume all energy within a restricted daily time period, appears to offer more sustainable weight loss and cardiometabolic changes and may be more acceptable as a permanent lifestyle change.

Eight hour TRF may have beneficial effects on improving menstruation, hyperandrogenemia and reducing weight especially body fat, decreasing insulin resistance and chronic inflammation in women with anovulatory PCOS. TRF may be suitable for PCOS women with appropriate counseling and patient management.

The progressive resistance training (PRT) improved hyperandrogenism and the menstrual cycle as well as the functional capacity with increased muscle strength and resulted in changes in body composition with increased lean muscle mass and decreased central obesity without a reduced total weight. There were also improvements in quality of life and sexual function as complementary benefits.

So, This study will be carried out in an attempt to know Which is more effective, Intermittent fasting diet or resistive exercise program on insulin resistance in obese woman with polycystic ovarian syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Seventy two obese women diagnosed with Polycystic ovarian syndrome by the gynecologist (based on the Rotterdam diagnostic criteria)
* Their age will range from 25 to 40 years old.
* Overweight or obese (BMI >25 kg/m2 and < 30 kg/m2).

Exclusion Criteria:

* The presence of diseases (such as congenital adrenal hyperplasia, Cushing syndrome, androgen secreting tumors, hyperprolactinemia, diabetes, thyroid diseases, Severe serious cardiovascular, gastrointestinal, kidney and liver diseases. premature ovarian failure, hypothalamic/pituitary disease
* Hormonal contraceptive use.
* Participants who did not complete the study were excluded from the analysis.
* Use of medication therapy that impacts carbohydrate or lipid metabolism (oral contraceptive pills, insulin sensitizers, anti epileptics, anti psychotics, statins, and fish oil) in the recent 6 months;
* Body weight fluctuations for more than 5% in the past 3 months; in preparation for pregnancy.
* Perimenopausal; night shift workers; fasting for more than 16 h per day; hypotension
* Alcohol intake for more than 100 g per week; smoking within the past 3 months
* Engaging in high intensity exercise.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
HOM-IR calculation | 8 weeks
  It is calculated from fasting glucose and fasting insulin. Different studies provide slightly different ranges for HOM-IR. But they all agree that the higher HOM-IR gets , the more insulin resistance are.
  Less than 1 : optimal insulin resistance. Above 1.9 : early insulin resistance. Above 2.9 : significant insulin resistance.

SECONDARY OUTCOMES:
Waist circumference measurement | 8 weeks
  It will be taken around the abdomen at the level of the umbilicus to measure waist circumference correctly. This will be performed before and after treatment for all groups (A,B and C).
Waist/ hip ratio assessment | 8 weeks
  It will be calculated as waist circumference in centimeters divided by hip circumference in centimeters. This will be performed before and after treatment for all groups (A,B and C).
Weight measurement | 8 weeks
  It will be measured before and after treatment for all groups (A,B and C), using the InBody GS 6.5 B.
Body mass index (BMI) measurement | 8 weeks
  It will be measured before and after treatment for all groups (A,B and C). The BMI will be calculated by the weight in kilograms divided by square of the height in centimeters according to the formula: BMI = weight (kg)/height2 (m2).
Body fat mass (BFM) measurement | 8 weeks
  It will be measured in kilogram before and after treatment for all groups (A,B and C), using the InBody GS 6.5 B.
Skeletal muscle mass (SMM) measurement | 8 weeks
  It will be measured in kilogram before and after treatment for all groups (A,B and C), using the InBody GS 6.5 B.

CONTACTS AND LOCATIONS:
Overall Officials: Soheir Mahmoud Elkosery, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Mashtoul Elsouq general Hospital, ‘Ezbet el-Sharika el-Miṣrîya, Egypt